CLINICAL TRIAL: NCT06751121
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWP14012-based Triple Therapy in Eradication of Helicobacter Pylori
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012-based Triple Therapy in Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012310
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Infected Patients; Helicobacter Pylori Infected Subjects
MeSH Terms: interventions — fexuprazan; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP14012 40 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg (Experimental): 1 tablet of DWP14012 40 mg + 1 capsule of DWC202301 30 mg placebo + amoxicillin 1000 mg (2 capsules of 500 mg) + 1 tablet of clarithromycin 500 mg
  Interventions: Drug: DWP14012 40mg; Drug: Amoxicillin 1000mg; Drug: Clarithromycin 500mg; Drug: DWC202301 30mg placebo
- DWC202301 30 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg (Active Comparator): 1 tablet of DWP14012 40 mg placebo + 1 capsule of DWC202301 30 mg + amoxicillin 1000 mg (2 capsules of 500 mg) + 1 tablet of clarithromycin 500 mg
  Interventions: Drug: DWC202301 30mg; Drug: Amoxicillin 1000mg; Drug: Clarithromycin 500mg; Drug: DWP14012 40mg placebo

INTERVENTIONS:
Drug: DWP14012 40mg — DWP14012 40 mg, tablet, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days).
  Arms: DWP14012 40 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg
Drug: DWC202301 30mg — DWC202301 30 mg, capsule, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days).
  Arms: DWC202301 30 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg
Drug: Amoxicillin 1000mg — Amoxicillin 1000 mg(2 capsules of 500mg), capsule, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days).
Drug: Clarithromycin 500mg — Clarithromycin 500 mg, tablet, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days)
Drug: DWC202301 30mg placebo — DWC202301 30 mg placebo, capsule, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days)
  Arms: DWP14012 40 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg
Drug: DWP14012 40mg placebo — DWP14012 40 mg placebo, tablet, orally, twice daily before a meal with the concomitant medications at the same time each day, if possible, during the treatment period (14 days)
  Arms: DWC202301 30 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg

SUMMARY:
This study is designed to demonstrate the non-inferiority and verify the safety of DWP14012-based triple therapy compared to DWC202301-based triple therapy as the first-line eradication therapy in patients who are positive for Helicobacter pylori

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females ≥19 and ≤75 years of age at the time of giving informed consent
2. Those who have all positive test results for H. pylori (13C-urea breath test and CLO) at screening visit (Visit 1)

   * A positive 13C-UBT result
   * A positive CLO result
3. Those who require treatment for H. pylori eradication as at least one of the following applies:

   * Those who have peptic ulcer (gastric ulcer or duodenal ulcer) based on an upper gastrointestinal (GI) endoscopy at screening visit (Visit 1)
   * Those who have chronic atrophic gastritis based on an upper GI endoscopy at screening visit (Visit 1)
   * Those with a history of endoscopic resection of early gastric cancer or gastric adenoma

Exclusion Criteria:

1. Those with significant upper GI bleeding
2. Those with a history of a surgical procedure that might affect gastric acid secretion (upper GI resection or vagotomy), or who are scheduled to undergo such procedure during this study
3. Those with Zollinger-Ellison syndrome or other gastric acid hypersecretion disorders
4. Those with a history of treatment for H. pylori eradication
5. Those with a history of any malignancy within recent 5 years prior to screening visit (Visit 1)

   * However, they can participate if 5 years have passed without recurrence after determined to achieve a complete remission (the complete removal of tumors through surgical procedures or the end of anticancer therapy)
   * Still, those with a history of malignancies in the digestive system, except early gastric cancer under the inclusion criteria, are excluded irrespective of a complete remission
6. Those who have experienced acute coronary artery disease (unstable angina, myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention), peripheral arterial disease and cerebrovascular disease (transient ischemic attack, stroke) within 24 weeks prior to screening visit (Visit 1)
7. Those with clinically significant systemic bleeding disorders, coagulation disorders, or severe blood disorders that make them ineligible for participation in this study
8. Those with acquired immunodeficiency syndrome (AIDS) or viral hepatitis (tested positive for HBs antigen or HCV antibody) (However, subjects who are negative for HCV-RNA can participate.)
9. Those who meet the following criteria according to the results of the hepatic or renal level test performed at screening visit (Visit 1)

   * At least one of ALT, AST, ALP, γ-GTP and total bilirubin > 2 times the upper limit of normal
   * BUN > 2 times the upper limit of normal
   * Creatinine clearance (CrCl) ≤ 30 mL/min
10. Patients with uncontrolled hypertension (systolic blood pressure of ≥ 160 mmHg or diastolic blood pressure of ≥ 100 mmHg at screening)
11. Patients with uncontrolled diabetes (HbA1c > 9.0 % at screening)
12. Patients with one or more of the following:

    * Heart failure (NYHA Class III ~ IV)
    * History of QT prolongation or ventricular arrhythmias (including Torsades de pointes)
13. Patients with hypokalemia (Potassium < 3 mmol/L at screening)
14. Patients with hypomagnesemia (Magnesium < 1.2 mg/dL at screening)
15. Those with clinically significant mental disorders
16. Patients with central nervous system infection
17. Patients with infectious mononucleosis
18. Those with a history of drug or alcohol abuse within recent 1 year prior to screening visit (Visit 1)
19. Those with a history of hypersensitivity or allergy to the IP, amoxicillin, clarithromycin, drugs used for 13C-UBT, or premedications for an upper GI endoscopy, or their components
20. Those with a history of hypersensitivity or allergy to proton pump inhibitors (PPIs), potassium-competitive acid blockers (P-CABs), benzimidazoles, penicillin antibiotics, or macrolide antibiotics
21. Those who are taking, or need to take, at least one of the following:

    * Atazanavir, Rilpivirine, or drugs that contain any of them
    * Pimozide, Domperidone
    * Ergot alkaloid and its derivatives (Ergotamine, Dihydroergotamine, etc.)
    * Mizolastine
    * Ticagrelor
    * Colchicine
22. Those who have a history of use of any PPIs, P-CABs or H2-receptor antagonists within recent 14 days prior to 13C-UBT of screening visit (Visit 1), or who need to take any of them during the study
23. Those who have a history of use of bismuth or any antibiotics known to be effective at eradication of H. pylori within recent 28 days prior to 13C-UBT of screening visit (Visit 1), or who need to take any of them during the study
24. For those using antibiotic resistance test results or samples prior to the screening visit (Visit 1), the subjects who have a history of antibiotic use from the time the results or samples were obtained (up to 90 days prior to the screening visit)
25. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
26. Those to whom an upper GI endoscopy cannot be performed
27. Pregnant or lactating women
28. Those who do not agree to use a proper contraception throughout the study duration

    * Proper contraception methods for the subject or his/her partner
    * Sterilization (vasectomy, etc.), or intrauterine devices (copper loop, intrauterine systems containing hormones)
    * Combined use of barrier methods with any one of non-oral hormonal contraceptives or spermicides
    * Combined use of a cervical cap or contraceptive diaphragm with male condoms
29. Those who have participated in other studies, and have been treated with the IP or medical device at least once within 4 weeks prior to participating in this study
30. Those deemed ineligible to participate in this study based on the investigator's other medical opinions

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | after at least 4 weeks (28 - 56 days) from the end of treatment
  H. pylori eradication rate identified by 13C-UBT after at least 4 weeks (28 - 56 days) from the end of treatment

SECONDARY OUTCOMES:
H. pylori eradication rate(for subjects who are resistant to clarithromycin) | after at least 4 weeks (28 - 56 days) from the end of treatment
  H. pylori eradication rate identified by 13C-UBT after at least 4 weeks (28 - 56 days) from the end of treatment (for subjects who are resistant to clarithromycin)
H. pylori eradication rate(for subjects who are not resistant to clarithromycin or amoxicillin) | after at least 4 weeks (28- 56 days) from the end of treatment
  H. pylori eradication rate identified by 13C-UBT after at least 4 weeks (28- 56 days) from the end of treatment (for subjects who are not resistant to clarithromycin or amoxicillin)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No